CLINICAL TRIAL: NCT01943461
Title: A Phase I Trial to Investigate the Tolerability, Safety, Pharmacokinetics, Biological and Clinical Activity of Avelumab (MSB0010718C) in Japanese Subjects With Metastatic or Locally Advanced Solid Tumors, With Expansion Part in Asian Subjects With Gastric Cancer
Brief Title: Avelumab in Metastatic or Locally Advanced Solid Tumors (JAVELIN Solid Tumor JPN)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: EMR 100070-002
Record Dates: First submitted 2013-09-06; First posted 2013-09-17 (Estimated); Results first posted 2020-09-30 (Actual); Last update posted 2020-09-30 (Actual); Status verified 2020-09

CONDITIONS: Solid Tumors
Keywords: Solid Tumors; MSB0010718C; anti PD-L1; avelumab; Phase 1
MeSH Terms: interventions — avelumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Dose-escalation Cohort: Avelumab 3 mg/kg (Experimental)
  Interventions: Drug: Avelumab 3 mg/kg
- Dose-escalation Cohort: Avelumab 10 mg/kg (Experimental)
  Interventions: Drug: Avelumab 10 mg/kg
- Dose-escalation Cohort: Avelumab 20 mg/kg (Experimental)
  Interventions: Drug: Avelumab 20 mg/kg
- Expansion Cohort: Avelumab 10 mg/kg (Experimental)
  Interventions: Drug: Avelumab 10 mg/kg

INTERVENTIONS:
Drug: Avelumab 3 mg/kg — Participants received intravenous infusion of Avelumab over 1 hour duration at a dose of 3 milligrams per kilogram (mg/kg) once every 2 weeks in the dose- escalation cohort until disease progression, unacceptable toxicity or withdrawal from the study or study drug occurred.
  Other Names: anti PD-L1; MSB0010718C
  Arms: Dose-escalation Cohort: Avelumab 3 mg/kg
Drug: Avelumab 10 mg/kg — Participants received intravenous infusion of Avelumab over 1 hour duration at a dose of 10 mg/kg once every 2 weeks in the dose- escalation cohort and expansion cohort until disease progression, unacceptable toxicity or withdrawal from the study or study drug occurred.
  Arms: Dose-escalation Cohort: Avelumab 10 mg/kg; Expansion Cohort: Avelumab 10 mg/kg
Drug: Avelumab 20 mg/kg — Participants received intravenous infusion of Avelumab over 1 hour duration at a dose of 20 mg/kg once every 2 weeks in the dose- escalation cohort until disease progression, unacceptable toxicity or withdrawal from the study or study drug occurred.
  Arms: Dose-escalation Cohort: Avelumab 20 mg/kg

SUMMARY:
This was a Phase 1, open-label, dose-escalation trial of avelumab (antibody targeting programmed death ligand 1 [anti PD-L1]) in Japanese participants with metastatic or locally advanced solid tumors, followed by a consecutive expansion part in Asian participants with gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent
* Male or female participants aged greater than or equal to (>=) 20 years
* For dose escalation part: Histologically or cytologically proven metastatic or locally advanced solid tumors, for which no standard therapy exists or standard therapy has failed
* For expansion part:

  * Availability of fresh and archive tumor in formalin fixed paraffin embedded tissue
  * With histologically or cytologically confirmed recurrent or refractory unresectable Stage IV gastric or gastro-esophageal junctional adenocarcinoma (according to American Joint Committee on Cancer/Union Internationale Contre le Cancer [UICC] 7th edition) and whose disease progressed after one or two prior chemotherapy regimen(s) involving both fluoropyrimidines and platinum
  * Presence of at least 1 measurable lesion according to RECIST version 1.1
  * Participants should not have severe peritoneal metastases. The following criteria were applied:

    * No clinical ileus or subileus
    * No moderate-to-severe ascites (participants with ascites restricted to the perihepatic space or pelvic cavity)
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1 at the trial entry and an estimated life expectancy of at least 3 months
* Adequate hematological, hepatic and renal function as defined in the protocol
* All participants must agree to use effective means of contraception with their partner from entry into the trial through 6 months after the last dose of avelumab

Exclusion Criteria:

* Concurrent treatment with a non-permitted drug
* Prior therapy with any antibody/drug targeting T cell co-regulatory proteins (immune checkpoints)
* Concurrent anticancer treatment or concurrent systemic therapy with steroids or other immunosuppressive agents, or use of any investigational drug within 30 days before the start of trial treatment. Short-term administration of steroids (that is, for allergic reactions or the management of immune-related adverse events [irAE]) is allowed
* Previous malignant disease within the last 5 years with the exception of adequately treated non-melanoma skin cancer, in situ cancer, or other cancer
* Non-oncology vaccine therapies for prevention of infection disease (e.g. seasonal flu vaccine, human papilloma virus vaccine) within 4 weeks of study drug administration. Vaccination while on study is also prohibited except for administration of the inactivated influenza vaccine.
* Pregnancy or lactation period
* Known alcohol or drug abuse
* Clinically significant (that is, active) cardiovascular disease
* All other significant diseases (for example, inflammatory bowel disease), which, in the opinion of the investigator, might impair the participant's tolerance of trial treatment
* Any psychiatric condition that would prohibit the understanding or rendering of informed consent
* Legal incapacity or limited legal capacity
* Other protocol defined exclusion criteria could apply

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2013-09-02 (Actual); Primary Completion 2015-01-07 (Actual); Study Completion 2019-09-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck KGaA, Darmstadt, Germany
Locations (1):
- Research site, Darmstadt, Germany

REFERENCES:
- [Background] Doi T, Iwasa S, Muro K, Satoh T, Hironaka S, Esaki T, Nishina T, Hara H, Machida N, Komatsu Y, Shimada Y, Otsu S, Shimizu S, Watanabe M. Phase 1 trial of avelumab (anti-PD-L1) in Japanese patients with advanced solid tumors, including dose expansion in patients with gastric or gastroesophageal junction cancer: the JAVELIN Solid Tumor JPN trial. Gastric Cancer. 2019 Jul;22(4):817-827. doi: 10.1007/s10120-018-0903-1. Epub 2018 Dec 4. PMID 30515672
- [Derived] Novakovic AM, Wilkins JJ, Dai H, Wade JR, Neuteboom B, Brar S, Bello CL, Girard P, Khandelwal A. Changing Body Weight-Based Dosing to a Flat Dose for Avelumab in Metastatic Merkel Cell and Advanced Urothelial Carcinoma. Clin Pharmacol Ther. 2020 Mar;107(3):588-596. doi: 10.1002/cpt.1645. Epub 2019 Nov 18. PMID 31553054
- See also: Trial Awareness and Transparency website — https://clinicaltrials.emdgroup.com/en/trial-details/?id=EMR100070-002
- See also: Medical Information Location Map - Med Info Contacts — http://www.merckgroup.com/en/company/contact-us/medinfo-contact-map.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Dose-escalation Cohort: Avelumab 3 mg/kg: Participants received intravenous infusion of Avelumab over 1 hour duration at a dose of 3 milligrams per kilogram (mg/kg) once every 2 weeks in the dose-escalation cohort until disease progression, unacceptable toxicity or withdrawal from the study or study drug occurred.
- Dose-escalation Cohort: Avelumab 10 mg/kg: Participants received intravenous infusion of Avelumab over 1 hour duration at a dose of 10 mg/kg once every 2 weeks in the dose-escalation cohort until disease progression, unacceptable toxicity or withdrawal from the study or study drug occurred.
- Dose-escalation Cohort: Avelumab 20 mg/kg: Participants received intravenous infusion of Avelumab over 1 hour duration at a dose of 20 mg/kg once every 2 weeks in the dose-escalation cohort until disease progression, unacceptable toxicity or withdrawal from the study or study drug occurred.
- Expansion Cohort: Avelumab 10 mg/kg: Participants received intravenous infusion of Avelumab over 1 hour duration at a dose of 10 mg/kg once every 2 weeks in the expansion cohort until disease progression, unacceptable toxicity or withdrawal from the study or study drug occurred.
Period: Overall Study
Arm/Group | Dose-escalation Cohort: Avelumab 3 mg/kg | Dose-escalation Cohort: Avelumab 10 mg/kg | Dose-escalation Cohort: Avelumab 20 mg/kg | Expansion Cohort: Avelumab 10 mg/kg
Started | 5 | 6 | 6 | 40
Completed | 5 | 6 | 6 | 40
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all participants who have received at least 1 dose of study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose-escalation Cohort: Avelumab 3 mg/kg | Dose-escalation Cohort: Avelumab 10 mg/kg | Dose-escalation Cohort: Avelumab 20 mg/kg | Expansion Cohort: Avelumab 10 mg/kg | Total
Number analyzed (Participants) | 5 | 6 | 6 | 40 | 57
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 5 | 2 | 22 | 32
  >=65 years | 2 | 1 | 4 | 18 | 25
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 3 | 11 | 18
  Male | 3 | 4 | 3 | 29 | 39
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 5 | 6 | 6 | 40 | 57
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 5 | 6 | 6 | 40 | 57
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Dose-escalation Cohorts: Number of Participants With Dose Limiting Toxicities (DLTs)
Description: DLT: any Grade greater than or equal to (>=) 3 or Adverse Events (AE) according to National Cancer Institute Common Toxicity Criteria for AE Version 4.03 (NCI-CTCAE v4.03); observed during first 3 weeks of dose-escalation part and as being related to Avelumab by Investigator/Sponsor. Following events were not considered as DLT: Grade 3 infusion-related reaction resolving to (<=) Grade 1 within 6 hours and controlled with medical management; Transient (<=6 hours) Grade 3 flulike symptoms/fever controlled with medical management and resolved to <= Grade 1;Transient (<=24 hours) Grade 3 fatigue, local reactions, headache, nausea, emesis that resolved to <=Grade1 with/without medical management, Grade 3 diarrhea, Grade 3 skin toxicity, Grade3 out-of-range laboratory values without any clinical correlate that resolves to <= Grade 1 or Baseline in < 7 days after medical management; Tumor flare phenomenon defined as local pain, irritation, rash localized at sites of known or suspected tumor.
Time Frame: Baseline up to 3 weeks
Population: DLT analysis set included all participants with data used for implementing the dose-escalation schedule.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose-escalation Cohort: Avelumab 3 mg/kg | Dose-escalation Cohort: Avelumab 10 mg/kg | Dose-escalation Cohort: Avelumab 20 mg/kg
Number analyzed (Participants) | 3 | 6 | 6
Participants | 0 | 0 | 0

2. Secondary Outcome: Dose-escalation Cohorts: Area Under the Serum Concentration-Time Curve From the Time of Dosing to the Time of the Last Observation (AUC0-t) of Avelumab
Description: Area under the serum concentration vs time curve from time zero to the last sampling time t at which the concentration was at or above the lower limit of quantification (LLOQ). AUC0-t was calculated by linear trapezoidal summation.
Time Frame: Within 6 hours before the infusion, at end of 1-hour infusion (Day 1), 0.5, 1, 2, 4, 6,12, 24, 36, 48, 168 hours after end of infusion
Population: Pharmacokinetic (PK) analysis set included all participants who have received at least 1 dose of study treatment and provided at least 1 measurable post-dose concentration.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*microgram per milliliter(hr*mcg/mL)
Arm/Group | Dose-escalation Cohort: Avelumab 3 mg/kg | Dose-escalation Cohort: Avelumab 10 mg/kg | Dose-escalation Cohort: Avelumab 20 mg/kg
Number analyzed (Participants) | 5 | 6 | 6
hour*microgram per milliliter(hr*mcg/mL) | 5120 (32.5) | 20100 (40.0) | 46800 (23.1)

3. Secondary Outcome: Dose-escalation Cohorts: Area Under the Serum Concentration-Time Curve From Time Zero Extrapolated to Infinity (AUC0-inf) of Avelumab
Description: Area under the curve from the time of dosing extrapolated to infinity was calculated by the linear trapezoidal summation and extrapolated to infinity using Clast/Lambda z after the first intravenous infusion. "Clast" was the last quantifiable concentration and "Lambda z" was terminal elimination rate constant determined by log-linear regression analysis of the measured serum concentrations of the terminal log-linear phase.
Time Frame: as for outcome 2
Population: PK analysis set included all participants who have received at least 1 dose of study treatment and provided at least 1 measurable post-dose concentration.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*mcg/mL
Arm/Group | Dose-escalation Cohort: Avelumab 3 mg/kg | Dose-escalation Cohort: Avelumab 10 mg/kg | Dose-escalation Cohort: Avelumab 20 mg/kg
Number analyzed (Participants) | 5 | 6 | 6
hr*mcg/mL | 6040 (27.5) | 24000 (47.4) | 53700 (24.3)

4. Secondary Outcome: Dose-escalation Cohorts: Maximum Observed Serum Concentration (Cmax) of Avelumab
Description: Cmax was obtained directly from the concentration versus time curve.
Time Frame: as for outcome 2
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg/mL
Arm/Group | Dose-escalation Cohort: Avelumab 3 mg/kg | Dose-escalation Cohort: Avelumab 10 mg/kg | Dose-escalation Cohort: Avelumab 20 mg/kg
Number analyzed (Participants) | 5 | 6 | 6
mcg/mL | 64 (22.2) | 179 (19.6) | 459 (13.6)

5. Secondary Outcome: Dose-escalation Cohorts: Time to Reach Maximum Observed Serum Concentration (Tmax) of Avelumab
Description: Tmax was time to reach maximum observed serum concentration obtained directly from the concentration versus time curve.
Time Frame: as for outcome 2
Population: as for outcome 3
Measure: Median (Full Range); unit: hour
Arm/Group | Dose-escalation Cohort: Avelumab 3 mg/kg | Dose-escalation Cohort: Avelumab 10 mg/kg | Dose-escalation Cohort: Avelumab 20 mg/kg
Number analyzed (Participants) | 5 | 6 | 6
hour | 1.683 [0.97 to 2.07] | 1.533 [1.00 to 3.08] | 1.683 [1.00 to 4.92]

6. Secondary Outcome: Dose-escalation Cohorts: Terminal Half-Life (t1/2) of Avelumab
Description: t1/2 was the time measured for the concentration to decrease by one half, determined as 0.693/Lambda z, here Lambda z was the terminal elimination rate constant determined by log-linear regression analysis of the measured serum concentrations of the terminal log-linear phase.
Time Frame: as for outcome 2
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour
Arm/Group | Dose-escalation Cohort: Avelumab 3 mg/kg | Dose-escalation Cohort: Avelumab 10 mg/kg | Dose-escalation Cohort: Avelumab 20 mg/kg
Number analyzed (Participants) | 5 | 6 | 6
hour | 94 (31.7) | 122 (33.1) | 112 (11.6)

7. Secondary Outcome: Dose-escalation Cohorts: Terminal Elimination Rate Constant (Lambda z) of Avelumab
Description: Terminal elimination rate constant was determined by log-linear regression analysis of the measured serum concentrations of the terminal log-linear phase. Participant wise data was reported for this outcome measure.
Time Frame: as for outcome 2
Population: PK analysis set included all participants who have received at least 1 dose of study treatment and provided at least 1 measurable post-dose concentration. The summarized data was not available for these arms therefore individual data was presented. Here, "Number Analyzed" signifies specific participant evaluated in respective arm.
Measure: Number; unit: per hour
Arm/Group | Dose-escalation Cohort: Avelumab 3 mg/kg | Dose-escalation Cohort: Avelumab 10 mg/kg | Dose-escalation Cohort: Avelumab 20 mg/kg
Number analyzed (Participants) | 5 | 6 | 6
per hour
  Participant 1: number analyzed (Participants) | 1 | 1 | 1
  Participant 1 | 0.00667 | 0.0103 | 0.00568
  Participant 2: number analyzed (Participants) | 1 | 1 | 1
  Participant 2 | 0.0114 | 0.00456 | 0.00750
  Participant 3: number analyzed (Participants) | 1 | 1 | 1
  Participant 3 | 0.00868 | 0.00456 | 0.00604
  Participant 4: number analyzed (Participants) | 1 | 1 | 1
  Participant 4 | 0.00663 | 0.00508 | 0.00568
  Participant 5: number analyzed (Participants) | 1 | 1 | 1
  Participant 5 | 0.00501 | 0.00476 | 0.00666
  Participant 6: number analyzed (Participants) | 0 | 1 | 1
  Participant 6 |  | 0.00662 | 0.00562

8. Secondary Outcome: Dose-escalation Cohorts: Programmed Death Ligand 1 (PD-L1) Receptor Occupancy
Description: Percentage of PD-L1 receptors occupied by avelumab on human lymphocytes (CD3+ cells) was assessed by flow cytometry on peripheral blood mononuclear cell (PBMC) samples. Greater than or equal to [>=] 85 percent [%] of cell viability was required for reliable receptor occupancy assessment.
Time Frame: Pre-infusion on Day 1; 4 and 48 hours after infusion on Day 3; Pre-infusion on Days 15, 29, 43, and 85
Population: Safety analysis set included all participants who have received at least 1 dose of study treatment.
Measure: Mean (Standard Deviation); unit: percentage of receptors
Arm/Group | Dose-escalation Cohort: Avelumab 3 mg/kg | Dose-escalation Cohort: Avelumab 10 mg/kg | Dose-escalation Cohort: Avelumab 20 mg/kg
Number analyzed (Participants) | 5 | 6 | 6
percentage of receptors | NA (NA) — Data could not analyzed because the analysis criterion was not met as all the PBMCs collected in the study had viability less than 85%. | NA (NA) — Data could not analyzed because the analysis criterion was not met as all the PBMCs collected in the study had viability less than 85%. | NA (NA) — Data could not analyzed because the analysis criterion was not met as all the PBMCs collected in the study had viability less than 85%.

9. Secondary Outcome: Dose-escalation Cohorts: Absolute Value of Cytokine Levels
Description: Cytokine analysis was performed to evaluate levels of Rantes, Monocyte chemoattractant protein-1 (MCP-1) and various interleukins (including IL-1 beta, IL-2, IL-4, IL-6, IL-10, IL-12p70, IL-13, IL-8), Tumor necrosis factors-alpha (TNF-alpha) and Interferon-gamma (IFN-gamma) in serum samples.
Time Frame: Day 1 (Pre-infusion), Day 3 (48 hours after infusion), Day 8 (168 hours after infusion), Day 15 (Pre-infusion), Day 43 (Pre-infusion), Day 45 (48 hours after infusion), Day 50 (168 hours after infusion)
Population: Safety analysis set included all participants who have received at least 1 dose of study treatment. Here "number analyzed" signified those participants who were evaluable for this outcome measure at the specified time points for the given category.
Measure: Mean (Standard Deviation); unit: nanogram per liter (ng/L)
Arm/Group | Dose-escalation Cohort: Avelumab 3 mg/kg | Dose-escalation Cohort: Avelumab 10 mg/kg | Dose-escalation Cohort: Avelumab 20 mg/kg
Number analyzed (Participants) | 5 | 6 | 6
nanogram per liter (ng/L)
  IFN-gamma: Day 1: Pre-Infusion | 9.094 (5.030) | 5.928 (4.331) | 7.723 (2.533)
  IFN-gamma: Day 3: 48 hours After Infusion | 17.716 (10.063) | 10.868 (3.609) | 18.810 (12.499)
  IFN-gamma: Day 8: 168 hours After Infusion | 15.016 (17.665) | 8.782 (3.118) | 12.198 (5.882)
  IFN-gamma: Day 15: Pre-Infusion | 21.347 (23.831) | 8.937 (2.557) | 17.998 (18.306)
  IFN-gamma: Day 43: Pre-Infusion: number analyzed (Participants) | 4 | 6 | 4
  IFN-gamma: Day 43: Pre-Infusion | 9.758 (3.838) | 15.947 (10.844) | 14.863 (13.232)
  IFN-gamma: Day 45: 48 hours After Infusion: number analyzed (Participants) | 4 | 6 | 4
  IFN-gamma: Day 45: 48 hours After Infusion | 21.153 (19.586) | 25.295 (28.939) | 41.253 (63.326)
  IFN-gamma: Day 50: 168 hours After Infusion: number analyzed (Participants) | 4 | 6 | 4
  IFN-gamma: Day 50: 168 hours After Infusion | 11.635 (6.705) | 16.503 (16.671) | 9.860 (4.818)
  IL-12P70: Day 1: Pre-Infusion | 0.200 (0.000) | 0.412 (0.401) | 0.200 (0.000)
  IL-12P70: Day 3: 48 hours After Infusion | 0.200 (0.000) | 0.395 (0.373) | 0.270 (0.171)
  IL-12P70: Day 8: 168 hours After Infusion | 0.200 (0.000) | 0.368 (0.412) | 0.237 (0.090)
  IL-12P70: Day 15: Pre- Infusion | 0.200 (0.000) | 0.395 (0.478) | 0.200 (0.000)
  IL-12P70: Day 43: Pre- Infusion: number analyzed (Participants) | 4 | 6 | 4
  IL-12P70: Day 43: Pre- Infusion | 0.200 (0.000) | 0.465 (0.375) | 0.200 (0.000)
  IL-12P70: Day 45: 48 hours After Infusion: number analyzed (Participants) | 4 | 6 | 4
  IL-12P70: Day 45: 48 hours After Infusion | 0.200 (0.000) | 0.447 (0.419) | 0.265 (0.130)
  IL-12P70: Day 50: 168 hours After Infusion: number analyzed (Participants) | 4 | 6 | 4
  IL-12P70: Day 50: 168 hours After Infusion | 0.200 (0.000) | 0.488 (0.479) | 0.348 (0.184)
  IL-10: Day 1: Pre-Infusion | 0.442 (0.470) | 0.504 (0.290) | 0.526 (0.401)
  IL-10: Day 3: 48 hours After Infusion | 0.768 (0.495) | 0.850 (0.506) | 0.960 (0.634)
  IL-10: Day 8: 168 hours After Infusion | 0.675 (0.680) | 0.993 (0.779) | 1.107 (0.805)
  IL-10: Day 15: Pre- Infusion | 0.686 (0.415) | 1.013 (0.838) | 1.045 (0.949)
  IL-10: Day 43: Pre -Infusion: number analyzed (Participants) | 4 | 6 | 4
  IL-10: Day 43: Pre -Infusion | 0.790 (0.770) | 2.098 (3.332) | 1.248 (1.495)
  IL-10: Day 45: 48 hours After Infusion: number analyzed (Participants) | 4 | 6 | 4
  IL-10: Day 45: 48 hours After Infusion | 1.574 (2.463) | 3.826 (7.268) | 2.185 (3.464)
  IL-10: Day 50:168 hours After Infusion: number analyzed (Participants) | 4 | 6 | 4
  IL-10: Day 50:168 hours After Infusion | 0.906 (1.227) | 2.199 (3.698) | 0.628 (0.411)
  IL-13: Day 1: Pre-Infusion | 0.540 (0.426) | 0.972 (0.230) | 1.430 (0.637)
  IL-13: Day 3: 48 hours After Infusion | 0.314 (0.165) | 0.995 (0.525) | 1.260 (0.890)
  IL-13: Day 8: 168 hours After Infusion | 0.684 (0.407) | 1.000 (0.372) | 1.052 (0.586)
  IL-13: Day 15: Pre- Infusion | 0.456 (0.301) | 1.073 (0.297) | 1.032 (0.564)
  IL-13: Day 43: Pre- Infusion: number analyzed (Participants) | 4 | 6 | 4
  IL-13: Day 43: Pre- Infusion | 0.508 (0.377) | 1.080 (0.513) | 1.453 (0.668)
  IL-13: Day 45: 48 hours After Infusion: number analyzed (Participants) | 4 | 6 | 4
  IL-13: Day 45: 48 hours After Infusion | 0.650 (0.398) | 0.840 (0.312) | 0.848 (0.469)
  IL-13: Day 50:168 hours After Infusion 4: number analyzed (Participants) | 4 | 6 | 4
  IL-13: Day 50:168 hours After Infusion 4 | 0.680 (0.344) | 0.910 (0.574) | 0.985 (0.534)
  IL-1beta: Day 1: Pre-Infusion | 0.255 (0.000) | 0.255 (0.000) | 0.255 (0.000)
  IL-1beta: Day 3: 48 hours After Infusion | 0.255 (0.000) | 0.255 (0.000) | 0.346 (0.222)
  IL-1beta: Day 8: 168 hours After Infusion | 0.255 (0.000) | 0.348 (0.227) | 0.255 (0.000)
  IL-1beta: Day 15: Pre- Infusion | 0.255 (0.000) | 0.255 (0.000) | 0.255 (0.000)
  IL-1beta: Day 43: Pre- Infusion: number analyzed (Participants) | 4 | 6 | 4
  IL-1beta: Day 43: Pre- Infusion | 0.255 (0.000) | 0.363 (0.263) | 0.255 (0.000)
  IL-1beta: Day 45: 48 hours After Infusion: number analyzed (Participants) | 4 | 6 | 4
  IL-1beta: Day 45: 48 hours After Infusion | 0.255 (0.000) | 0.543 (0.704) | 0.255 (0.000)
  IL-1beta: Day 50: 168 hours After Infusion: number analyzed (Participants) | 4 | 6 | 4
  IL-1beta: Day 50: 168 hours After Infusion | 0.255 (0.000) | 0.516 (0.639) | 0.255 (0.000)
  IL-2: Day 1: Pre-Infusion | 0.400 (0.220) | 0.452 (0.274) | 0.458 (0.472)
  IL-2: Day 3: 48 hours After Infusion | 0.396 (0.126) | 0.670 (0.334) | 0.608 (0.490)
  IL-2: Day 8: 168 hours After Infusion | 0.354 (0.162) | 0.475 (0.330) | 0.675 (0.886)
  IL-2: Day 15: Pre-Infusion | 0.320 (0.130) | 0.300 (0.209) | 0.417 (0.397)
  IL-2: Day 43: Pre- Infusion: number analyzed (Participants) | 4 | 6 | 4
  IL-2: Day 43: Pre- Infusion | 0.388 (0.148) | 0.500 (0.273) | 0.470 (0.362)
  IL-2: Day 45: 48 hours After Infusion: number analyzed (Participants) | 4 | 6 | 4
  IL-2: Day 45: 48 hours After Infusion | 0.438 (0.388) | 0.470 (0.345) | 0.488 (0.404)
  IL-2: Day 50: 168 hours After Infusion: number analyzed (Participants) | 4 | 6 | 4
  IL-2: Day 50: 168 hours After Infusion | 0.448 (0.241) | 0.465 (0.278) | 0.485 (0.411)
  IL-4: Day 1: Pre-Infusion | 0.100 (0.000) | 0.100 (0.000) | 0.100 (0.000)
  IL-4: Day 3: 48 hours After Infusion | 0.100 (0.000) | 0.100 (0.000) | 0.100 (0.000)
  IL-4: Day 8: 168 hours After Infusion | 0.100 (0.000) | 0.100 (0.000) | 0.130 (0.073)
  IL-4: Day 15: Pre-Infusion | 0.100 (0.000) | 0.100 (0.000) | 0.100 (0.000)
  IL-4: Day 43: Pre- Infusion: number analyzed (Participants) | 4 | 6 | 4
  IL-4: Day 43: Pre- Infusion | 0.100 (0.000) | 0.100 (0.000) | 0.100 (0.000)
  IL-4: Day 45: 48 hours After Infusion: number analyzed (Participants) | 4 | 6 | 4
  IL-4: Day 45: 48 hours After Infusion | 0.100 (0.000) | 0.100 (0.000) | 0.100 (0.000)
  IL-4: Day 50: 168 hours After Infusion: number analyzed (Participants) | 4 | 6 | 4
  IL-4: Day 50: 168 hours After Infusion | 0.100 (0.000) | 0.100 (0.000) | 0.100 (0.000)
  IL-6: Day 1: Pre-Infusion | 1.372 (0.917) | 3.633 (6.078) | 1.245 (0.238)
  IL-6: Day 3: 48 hours After Infusion | 1.398 (0.713) | 3.843 (5.018) | 6.433 (11.449)
  IL-6: Day 8: 168 hours After Infusion | 1.740 (1.270) | 2.922 (3.538) | 1.788 (0.529)
  IL-6: Day 15: Pre- Infusion | 2.032 (2.620) | 3.325 (2.939) | 1.890 (1.097)
  IL-6: Day 43: Pre- Infusion: number analyzed (Participants) | 4 | 6 | 4
  IL-6: Day 43: Pre- Infusion | 2.215 (3.279) | 1.978 (2.070) | 2.995 (2.500)
  IL-6: Day 45: 48 hours After Infusion: number analyzed (Participants) | 4 | 6 | 4
  IL-6: Day 45: 48 hours After Infusion | 2.888 (4.548) | 3.583 (6.013) | 3.065 (2.355)
  IL-6: Day 50: 168 hours After Infusion: number analyzed (Participants) | 4 | 6 | 4
  IL-6: Day 50: 168 hours After Infusion | 1.468 (1.544) | 4.082 (6.986) | 5.533 (4.287)
  MCP-1: Day 1: Pre-Infusion | 243.664 (55.976) | 209.280 (31.895) | 268.415 (52.240)
  MCP-1: Day 3: 48 hours After Infusion | 289.148 (69.117) | 250.230 (71.660) | 276.765 (30.402)
  MCP-1: Day 8: 168 hours After Infusion | 257.706 (69.318) | 229.240 (56.104) | 292.260 (47.383)
  MCP-1: Day 15: Pre- Infusion | 257.888 (93.740) | 226.445 (28.636) | 267.008 (38.395)
  MCP-1: Day 43: Pre- Infusion: number analyzed (Participants) | 4 | 6 | 4
  MCP-1: Day 43: Pre- Infusion | 282.053 (65.125) | 218.855 (45.141) | 228.460 (53.309)
  MCP-1: Day 45: 48 hours After Infusion | 258.265 (57.606) | 268.657 (84.748) | 235.265 (40.957)
  MCP-1: Day 50: 168 hours After Infusion: number analyzed (Participants) | 4 | 6 | 4
  MCP-1: Day 50: 168 hours After Infusion | 274.320 (49.826) | 241.980 (70.308) | 242.380 (15.451)
  Rantes: Day 1: Pre-Infusion: number analyzed (Participants) | 4 | 6 | 6
  Rantes: Day 1: Pre-Infusion | 32292.35 (24365.33) | 33583.68 (26542.38) | 35038.29 (6936.25)
  Rantes: Day 3: 48 hours After Infusion | 31514.77 (13931.92) | 54874.62 (45162.06) | 29282.41 (3512.35)
  Rantes: Day 8: 168 hours After Infusion | 36607.67 (19388.38) | 52933.35 (37662.84) | 28655.39 (8282.64)
  Rantes: Day 15: Pre-Infusion: number analyzed (Participants) | 4 | 6 | 4
  Rantes: Day 15: Pre-Infusion | 59985.74 (21964.23) | 45301.97 (19703.88) | 34758.15 (9429.32)
  Rantes: Day 43: Pre-Infusion: number analyzed (Participants) | 4 | 6 | 4
  Rantes: Day 43: Pre-Infusion | 30657.45 (6773.47) | 43532.09 (25175.05) | 36738.48 (10865.40)
  Rantes: Day 45: 48 hours After Infusion: number analyzed (Participants) | 4 | 6 | 4
  Rantes: Day 45: 48 hours After Infusion | 28777.63 (10267.15) | 41629.09 (25017.89) | 34107.87 (15731.50)
  Rantes: Day 50: 168 hours After Infusion: number analyzed (Participants) | 4 | 6 | 4
  Rantes: Day 50: 168 hours After Infusion | 38235.52 (6740.02) | 52287.81 (35615.67) | 41265.30 (9052.83)
  TNF-alpha: Day 1: Pre-Infusion | 2.304 (0.564) | 2.582 (0.986) | 2.188 (0.650)
  TNF-alpha: Day 3: 48 hours After Infusion | 3.482 (0.971) | 4.403 (1.578) | 3.607 (1.579)
  TNF-alpha: Day 8: 168 hours After Infusion | 2.440 (0.763) | 3.233 (1.174) | 2.682 (0.994)
  TNF-alpha: Day 15: Pre-Infusion | 2.832 (1.523) | 3.155 (1.154) | 2.720 (0.969)
  TNF-alpha: Day 43: Pre-Infusion: number analyzed (Participants) | 4 | 6 | 4
  TNF-alpha: Day 43: Pre-Infusion | 2.720 (0.908) | 3.490 (1.987) | 2.698 (1.063)
  TNF-alpha: Day 45: 48 hours After Infusion: number analyzed (Participants) | 4 | 6 | 4
  TNF-alpha: Day 45: 48 hours After Infusion | 3.983 (3.359) | 3.935 (2.316) | 3.218 (1.807)
  TNF-alpha: Day 50: 168 hours After Infusion: number analyzed (Participants) | 4 | 6 | 4
  TNF-alpha: Day 50: 168 hours After Infusion | 3.180 (2.200) | 3.967 (2.515) | 2.525 (0.965)
  IL-8: Day 1: Pre-Infusion | 23.210 (26.035) | 20.517 (7.254) | 31.667 (34.892)
  IL-8: Day 3: 48 hours After Infusion | 30.122 (28.378) | 31.717 (14.891) | 44.033 (42.682)
  IL-8: Day 8: 168 hours After Infusion | 31.082 (35.176) | 29.750 (20.021) | 36.500 (40.883)
  IL-8: Day 15: Pre- Infusion | 24.372 (25.645) | 23.817 (12.850) | 46.967 (68.781)
  IL-8: Day 43: Pre-Infusion: number analyzed (Participants) | 4 | 6 | 4
  IL-8: Day 43: Pre-Infusion | 56.310 (88.524) | 25.733 (14.433) | 17.600 (5.614)
  IL-8: Day 45: 48 hours After Infusion: number analyzed (Participants) | 4 | 6 | 4
  IL-8: Day 45: 48 hours After Infusion | 51.015 (74.760) | 30.083 (17.206) | 21.300 (7.806)
  IL-8: Day 50: 168 hours After Infusion: number analyzed (Participants) | 4 | 6 | 4
  IL-8: Day 50: 168 hours After Infusion | 65.448 (104.447) | 28.783 (11.963) | 19.028 (9.162)

10. Secondary Outcome: Dose-escalation Cohorts: Log Fold Change From Baseline in Cytokine Levels
Description: Cytokine analysis was performed to evaluate levels of Rantes, Monocyte chemoattractant protein-1 (MCP-1) and various interleukins (including IL-1beta, IL-2, IL-4, IL-6, IL-10, IL-12p70, IL-13, IL-8), Tumor necrosis factors-alpha (TNF-alpha) and Interferon-gamma (IFN-gamma) in serum samples. Log fold change from baseline (logFC) was defined as logFC (cytokine at time t) = log (cytokine signal at time t) - log (cytokine signal at baseline).
Time Frame: Baseline (Day 1 [Pre-infusion]), Day 3 (48 hours after infusion), Day 8 (168 hours after infusion), Day 15 (Pre-infusion), Day 43 (Pre-infusion), Day 45 (48 hours after infusion), Day 50 (168 hours after infusion)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: log fold change
Arm/Group | Dose-escalation Cohort: Avelumab 3 mg/kg | Dose-escalation Cohort: Avelumab 10 mg/kg | Dose-escalation Cohort: Avelumab 20 mg/kg
Number analyzed (Participants) | 5 | 6 | 6
log fold change
  IFN-gamma: Day 3: 48 hours After Infusion | 0.903 (1.258) | 1.038 (0.689) | 1.096 (0.975)
  IFN-gamma: Day 8: 168 hours After Infusion | 0.280 (1.365) | 0.722 (0.945) | 0.600 (0.243)
  IFN-gamma: Day 15: Pre-Infusion | 0.396 (1.958) | 0.779 (0.654) | 0.867 (0.690)
  IFN-gamma: Day 43: Pre-Infusion: number analyzed (Participants) | 4 | 6 | 4
  IFN-gamma: Day 43: Pre-Infusion | 0.071 (0.800) | 1.335 (1.735) | 0.631 (0.593)
  IFN-gamma: Day 45: 48 hours After Infusion: number analyzed (Participants) | 4 | 6 | 4
  IFN-gamma: Day 45: 48 hours After Infusion | 0.768 (1.925) | 1.617 (2.037) | 1.215 (1.576)
  IFN-gamma: Day 50: 168 hours After Infusion: number analyzed (Participants) | 4 | 6 | 4
  IFN-gamma: Day 50: 168 hours After Infusion | 0.234 (1.385) | 1.045 (2.010) | 0.273 (0.249)
  IL-12P70: Day 3: 48 hours After Infusion | 0.000 (0.000) | -0.030 (0.750) | 0.272 (0.666)
  IL-12P70: Day 8: 168 hours After Infusion | 0.000 (0.000) | -0.203 (0.504) | 0.178 (0.437)
  IL-12P70: Day 15: Pre- Infusion | 0.000 (0.000) | -0.174 (0.524) | 0.000 (0.000)
  IL-12P70: Day 43: Pre- Infusion: number analyzed (Participants) | 4 | 6 | 4
  IL-12P70: Day 43: Pre- Infusion | 0.000 (0.000) | 0.239 (0.990) | 0.000 (0.000)
  IL-12P70: Day 45: 48 hours After Infusion: number analyzed (Participants) | 4 | 6 | 4
  IL-12P70: Day 45: 48 hours After Infusion | 0.000 (0.000) | 0.087 (0.950) | 0.300 (0.601)
  IL-12P70: Day 50: 168 hours After Infusion: number analyzed (Participants) | 4 | 6 | 4
  IL-12P70: Day 50: 168 hours After Infusion | 0.000 (0.000) | 0.151 (1.033) | 0.643 (0.770)
  IL-10: Day 3: 48 hours After Infusion | 1.103 (0.888) | 0.743 (0.371) | 0.942 (0.199)
  IL-10: Day 8: 168 hours After Infusion | 0.624 (1.081) | 0.704 (0.962) | 1.088 (0.348)
  IL-10: Day 15: Pre- Infusion | 0.972 (0.691) | 0.720 (0.978) | 0.942 (0.444)
  IL-10: Day 43: Pre-Infusion: number analyzed (Participants) | 4 | 6 | 4
  IL-10: Day 43: Pre-Infusion | 0.919 (0.736) | 1.072 (1.452) | 1.317 (1.238)
  IL-10: Day 45: 48 hours After Infusion: number analyzed (Participants) | 4 | 6 | 4
  IL-10: Day 45: 48 hours After Infusion | 0.976 (1.416) | 1.375 (1.767) | 1.467 (1.758)
  IL-10: Day 50:168 hours After Infusion: number analyzed (Participants) | 4 | 6 | 4
  IL-10: Day 50:168 hours After Infusion | 0.633 (1.122) | 1.041 (1.680) | 0.761 (0.713)
  IL-13: Day 3: 48 hours After Infusion | -0.541 (0.980) | -0.170 (0.844) | -0.416 (1.245)
  IL-13: Day 8: 168 hours After Infusion | 0.407 (0.896) | -0.004 (0.245) | -0.581 (0.490)
  IL-13: Day 15: Pre- Infusion | -0.133 (1.191) | 0.125 (0.467) | -0.603 (0.519)
  IL-13: Day 43: Pre- Infusion: number analyzed (Participants) | 4 | 6 | 4
  IL-13: Day 43: Pre- Infusion | 0.353 (1.670) | -0.044 (0.866) | 0.200 (0.391)
  IL-13: Day 45: 48 hours After Infusion: number analyzed (Participants) | 4 | 6 | 4
  IL-13: Day 45: 48 hours After Infusion | 0.769 (1.778) | -0.327 (0.729) | -0.660 (0.560)
  IL-13: Day 50:168 hours After Infusion 4: number analyzed (Participants) | 4 | 6 | 4
  IL-13: Day 50:168 hours After Infusion 4 | 0.867 (1.796) | -0.427 (1.082) | -0.319 (0.615)
  IL-1beta: Day 3: 48 hours After Infusion | 0.000 (0.000) | 0.000 (0.000) | 0.275 (0.673)
  IL-1beta: Day 8: 168 hours After Infusion | 0.000 (0.000) | 0.278 (0.681) | 0.000 (0.000)
  IL-1beta: Day 15: Pre- Infusion | 0.000 (0.000) | 0.000 (0.000) | 0.000 (0.000)
  IL-1beta: Day 43: Pre-Infusion: number analyzed (Participants) | 4 | 6 | 4
  IL-1beta: Day 43: Pre-Infusion | 0.000 (0.000) | 0.303 (0.743) | 0.000 (0.000)
  IL-1beta: Day 45: 48 hours After Infusion: number analyzed (Participants) | 4 | 6 | 4
  IL-1beta: Day 45: 48 hours After Infusion | 0.000 (0.000) | 0.493 (1.207) | 0.000 (0.000)
  IL-1beta: Day 50: 168 hours After Infusion: number analyzed (Participants) | 4 | 6 | 4
  IL-1beta: Day 50: 168 hours After Infusion | 0.000 (0.000) | 0.473 (1.158) | 0.000 (0.000)
  IL-2: Day 3: 48 hours After Infusion | 0.108 (1.340) | 0.664 (0.749) | 0.531 (0.628)
  IL-2: Day 8: 168 hours After Infusion | -0.118 (1.230) | 0.035 (0.906) | 0.326 (0.545)
  IL-2: Day 15: Pre-Infusion | -0.228 (1.134) | -0.577 (1.055) | -0.059 (0.096)
  IL-2: Day 43: Pre- Infusion: number analyzed (Participants) | 4 | 6 | 4
  IL-2: Day 43: Pre- Infusion | 0.296 (1.375) | 0.211 (0.754) | -0.193 (0.243)
  IL-2: Day 45: 48 hours After Infusion: number analyzed (Participants) | 4 | 6 | 4
  IL-2: Day 45: 48 hours After Infusion | 0.194 (1.675) | 0.009 (0.892) | -0.175 (0.202)
  IL-2: Day 50: 168 hours After Infusion: number analyzed (Participants) | 4 | 6 | 4
  IL-2: Day 50: 168 hours After Infusion | 0.432 (1.547) | 0.099 (0.608) | -0.188 (0.220)
  IL-4: Day 3: 48 hours After Infusion | 0.000 (0.000) | 0.000 (0.000) | 0.000 (0.000)
  IL-4: Day 8: 168 hours After Infusion | 0.000 (0.000) | 0.000 (0.000) | 0.248 (0.606)
  IL-4: Day 15: Pre-Infusion | 0.000 (0.000) | 0.000 (0.000) | 0.000 (0.000)
  IL-4: Day 43: Pre- Infusion: number analyzed (Participants) | 4 | 6 | 4
  IL-4: Day 43: Pre- Infusion | 0.000 (0.000) | 0.000 (0.000) | 0.000 (0.000)
  IL-4: Day 45: 48 hours After Infusion: number analyzed (Participants) | 4 | 6 | 4
  IL-4: Day 45: 48 hours After Infusion | 0.000 (0.000) | 0.000 (0.000) | 0.000 (0.000)
  IL-4: Day 50: 168 hours After Infusion: number analyzed (Participants) | 4 | 6 | 4
  IL-4: Day 50: 168 hours After Infusion | 0.000 (0.000) | 0.000 (0.000) | 0.000 (0.000)
  IL-6: Day 3: 48 hours After Infusion | 0.153 (0.897) | 0.660 (0.816) | 1.196 (1.614)
  IL-6: Day 8: 168 hours After Infusion | 0.314 (0.421) | 0.194 (0.618) | 0.498 (0.321)
  IL-6: Day 15: Pre- Infusion | 0.069 (1.455) | 0.451 (1.457) | 0.474 (0.572)
  IL-6: Day 43: Pre- Infusion: number analyzed (Participants) | 4 | 6 | 4
  IL-6: Day 43: Pre- Infusion | 0.068 (0.949) | -0.009 (0.980) | 1.112 (0.898)
  IL-6: Day 45: 48 hours After Infusion: number analyzed (Participants) | 4 | 6 | 4
  IL-6: Day 45: 48 hours After Infusion | 0.273 (1.187) | 0.116 (0.676) | 1.158 (0.998)
  IL-6: Day 50: 168 hours After Infusion: number analyzed (Participants) | 4 | 6 | 4
  IL-6: Day 50: 168 hours After Infusion | 0.064 (0.573) | 0.279 (0.690) | 1.883 (1.287)
  MCP-1: Day 3: 48 hours After Infusion | 0.242 (0.206) | 0.213 (0.296) | 0.062 (0.234)
  MCP-1: Day 8: 168 hours After Infusion | 0.067 (0.278) | 0.110 (0.297) | 0.132 (0.202)
  MCP-1: Day 15: Pre- Infusion | -0.010 (0.684) | 0.120 (0.141) | 0.005 (0.211)
  MCP-1: Day 43: Pre- Infusion: number analyzed (Participants) | 4 | 6 | 4
  MCP-1: Day 43: Pre- Infusion | 0.173 (0.358) | 0.055 (0.343) | -0.232 (0.150)
  MCP-1: Day 45: 48 hours After Infusion: number analyzed (Participants) | 4 | 6 | 4
  MCP-1: Day 45: 48 hours After Infusion | 0.045 (0.209) | 0.318 (0.383) | -0.176 (0.183)
  MCP-1: Day 50: 168 hours After Infusion: number analyzed (Participants) | 4 | 6 | 4
  MCP-1: Day 50: 168 hours After Infusion | 0.144 (0.226) | 0.180 (0.394) | -0.118 (0.420)
  Rantes: Day 3: 48 hours After Infusion: number analyzed (Participants) | 4 | 6 | 6
  Rantes: Day 3: 48 hours After Infusion | 0.198 (0.849) | 0.589 (0.927) | -0.242 (0.383)
  Rantes: Day 8: 168 hours After Infusion: number analyzed (Participants) | 4 | 6 | 6
  Rantes: Day 8: 168 hours After Infusion | 0.289 (1.709) | 0.615 (0.866) | -0.325 (0.625)
  Rantes: Day 15: Pre-Infusion: number analyzed (Participants) | 3 | 6 | 6
  Rantes: Day 15: Pre-Infusion | 0.997 (1.992) | 0.582 (0.649) | -0.025 (0.360)
  Rantes: Day 43: Pre-Infusion: number analyzed (Participants) | 4 | 6 | 4
  Rantes: Day 43: Pre-Infusion | 0.389 (1.452) | 0.450 (0.765) | -0.079 (0.306)
  Rantes: Day 45: 48 hours After Infusion: number analyzed (Participants) | 4 | 6 | 4
  Rantes: Day 45: 48 hours After Infusion | 0.249 (1.947) | 0.353 (0.809) | -0.257 (0.487)
  Rantes: Day 50: 168 hours After Infusion: number analyzed (Participants) | 4 | 6 | 4
  Rantes: Day 50: 168 hours After Infusion | 0.718 (1.386) | 0.656 (0.634) | 0.107 (0.326)
  TNF-alpha: Day 3: 48 hours After Infusion | 0.589 (0.443) | 0.770 (0.314) | 0.646 (0.388)
  TNF-alpha: Day 8: 168 hours After Infusion | 0.065 (0.378) | 0.343 (0.195) | 0.262 (0.144)
  TNF-alpha: Day 15: Pre-Infusion | 0.182 (0.805) | 0.301 (0.090) | 0.292 (0.158)
  TNF-alpha: Day 43: Pre-Infusion: number analyzed (Participants) | 4 | 6 | 4
  TNF-alpha: Day 43: Pre-Infusion | 0.329 (0.253) | 0.365 (0.304) | 0.216 (0.184)
  TNF-alpha: Day 45: 48 hours After Infusion: number analyzed (Participants) | 4 | 6 | 4
  TNF-alpha: Day 45: 48 hours After Infusion | 0.612 (0.848) | 0.527 (0.376) | 0.382 (0.422)
  TNF-alpha: Day 50: 168 hours After Infusion: number analyzed (Participants) | 4 | 6 | 4
  TNF-alpha: Day 50: 168 hours After Infusion | 0.400 (0.672) | 0.507 (0.378) | 0.119 (0.134)
  IL-8: Day 3: 48 hours After Infusion | 0.604 (0.553) | 0.539 (0.400) | 0.554 (0.484)
  IL-8: Day 8: 168 hours After Infusion | 0.444 (0.313) | 0.393 (0.406) | 0.189 (0.145)
  IL-8: Day 15: Pre- Infusion | 0.201 (0.560) | 0.118 (0.467) | 0.256 (0.536)
  IL-8: Day 43: Pre-Infusion: number analyzed (Participants) | 4 | 6 | 4
  IL-8: Day 43: Pre-Infusion | 0.773 (1.073) | 0.241 (0.388) | 0.033 (0.367)
  IL-8: Day 45: 48 hours After Infusion: number analyzed (Participants) | 4 | 6 | 4
  IL-8: Day 45: 48 hours After Infusion | 0.858 (0.885) | 0.451 (0.330) | 0.283 (0.499)
  IL-8: Day 50: 168 hours After Infusion: number analyzed (Participants) | 4 | 6 | 4
  IL-8: Day 50: 168 hours After Infusion | 0.924 (1.088) | 0.441 (0.284) | 0.081 (0.798)

11. Secondary Outcome: Dose-escalation Cohorts: Number of Participants With Treatment-Emergent Positive Human Anti-Human Antibody (HAHA)
Description: Participants not having positive HAHA prior to treatment with Avelumab and with at least one positive post-baseline result in the HAHA assay were termed as treatment-emergent. Treatment-emergent participants were further classified as Transient Positive or Persistent positive. Participants were considered as transient positive if time between first and last positive result was less than 16 weeks apart and a negative result at the most recent visit. Participants were considered as persistent positive if time between first and last positive result greater than or equal to [>=] 16 weeks apart or a positive evaluation at the most recent visit. Number of participants with treatment-emergent positive HAHA were reported.
Time Frame: Day 15 up to Day 2205
Population: Safety analysis set included all participants who have received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose-escalation Cohort: Avelumab 3 mg/kg | Dose-escalation Cohort: Avelumab 10 mg/kg | Dose-escalation Cohort: Avelumab 20 mg/kg
Number analyzed (Participants) | 5 | 6 | 6
Participants
  Transient positive treatment emergent | 0 | 0 | 0
  Persistent positive treatment emergent | 1 | 0 | 0

12. Secondary Outcome: Dose-escalation Cohorts: Number of Participants With Treatment-Emergent Adverse Events (TEAEs), Serious TEAEs, TEAEs Leading to Death, and TEAEs Leading to Discontinuation
Description: An Adverse Event (AE) was defined as any unfavourable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of study drug, whether or not considered related to the study drug or worsening of pre-existing medical condition, whether or not related to study drug. A serious adverse event (SAE) was an AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect or was otherwise considered medically important. TEAEs were those events with onset dates occurring during the on-treatment period for the first time, or if the worsening of an event was during the on-treatment period. TEAEs included both serious TEAEs and non-serious TEAEs.
Time Frame: Time from first dose of study treatment up to 2205 days
Population: Safety analysis set included all participants who have received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose-escalation Cohort: Avelumab 3 mg/kg | Dose-escalation Cohort: Avelumab 10 mg/kg | Dose-escalation Cohort: Avelumab 20 mg/kg
Number analyzed (Participants) | 5 | 6 | 6
Participants
  TEAEs | 5 | 6 | 5
  Serious TEAEs | 1 | 0 | 2
  TEAEs Leading To Discontinuation | 0 | 0 | 1
  TEAEs Leading To Death | 1 | 0 | 0

13. Secondary Outcome: Expansion Cohort: Area Under the Serum Concentration-Time Curve From the Time of Dosing to the End of Dose Interval (AUC0-336hour [hr]) of Avelumab
Description: AUC0-336hour was defined as area under the serum concentration-time curve from the time of dosing to the end of dose interval (336 hr). It was calculated by linear trapezoidal summation.
Time Frame: Within 6 hours before and the end of the 1-hour infusion (Day 1) and 336 hours after end of infusion
Population: PK analysis set included all participants who have received at least 1 dose of study treatment and provided at least 1 measurable post-dose concentration. Here "Number of participants analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Expansion Cohort: Avelumab 10 mg/kg
Number analyzed (Participants) | 37
mcg/mL | 14.525 (6.3064)

14. Secondary Outcome: Expansion Cohort: Serum Trough Concentration Levels (Ctrough) of Avelumab
Description: Ctrough was defined as the trough or minimum serum concentration.
Time Frame: Within 6 hours before the 1-hour infusion on Day 15, Day 29, Day 43, Day 85, Day 127 and Day 169.
Population: PK analysis set: all participants who have received at least 1 dose of study treatment and provided at least 1 measurable post-dose concentration. "Overall Number of Participants Analyzed" = participants evaluable for this outcome measure and "Number analyzed" = participants who were evaluable at the specified time points for the given category.
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Expansion Cohort: Avelumab 10 mg/kg
Number analyzed (Participants) | 37
mcg/mL
  Day 15 | 14.525 (6.3064)
  Day 29: number analyzed (Participants) | 34
  Day 29 | 17.366 (9.2981)
  Day 43: number analyzed (Participants) | 28
  Day 43 | 19.686 (9.0747)
  Day 85: number analyzed (Participants) | 15
  Day 85 | 25.125 (14.4089)
  Day 127: number analyzed (Participants) | 9
  Day 127 | 22.544 (16.7706)
  Day 169: number analyzed (Participants) | 5
  Day 169 | 20.857 (23.2820)

15. Secondary Outcome: Expansion Cohort: Number of Participants With Programmed Death Ligand 1 (PD-L1) Tumor Expression
Description: The PD-L1 expression was evaluated using an established antiPD-L1 immunohistochemistry (IHC) assay.
Time Frame: Time from first dose of study treatment up to 1906 days
Population: Safety analysis set included all participants who have received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Expansion Cohort: Avelumab 10 mg/kg
Number analyzed (Participants) | 40
Participants | 11

16. Secondary Outcome: Expansion Cohort: Absolute Values of Cytokine Levels
Description: Cytokine analysis was performed to evaluate levels of Monocyte chemoattractant protein-1 (MCP-1) and various interleukins (including IL-5, IL-6, IL-8), Tumor necrosis factors-alpha (TNF-alpha) and Interferon-gamma (IFN-gamma) in serum samples.
Time Frame: Day 1 (Pre-infusion), Day 8 (168 hour after infusion) and Day 43 (Pre-infusion)
Population: Safety analysis set included all participants who have received at least 1 dose of study treatment. Here "Number Analyzed" = participants who were evaluable for this outcome measure at the specified time points for the given category.
Measure: Mean (Standard Deviation); unit: nanogram per liter (ng/L)
Arm/Group | Expansion Cohort: Avelumab 10 mg/kg
Number analyzed (Participants) | 40
nanogram per liter (ng/L)
  IFN-gamma: Day 1: Pre-Infusion | 28.125 (97.504)
  IFN-gamma: Day 8: 168 hours post Infusion | 23.063 (25.899)
  IFN-gamma: Day 43: Pre-Infusion: number analyzed (Participants) | 28
  IFN-gamma: Day 43: Pre-Infusion | 19.215 (22.041)
  IL-5: Day 1: Pre-Infusion | 1.139 (1.596)
  IL-5: Day 8: 168 hours Post Infusion | 1.492 (2.135)
  IL-5: Day 43: Pre-Infusion: number analyzed (Participants) | 28
  IL-5: Day 43: Pre-Infusion | 1.632 (1.958)
  IL-6: Day 1: Pre-Infusion | 3.502 (7.968)
  IL-6: Day 8: 168 hours Post Infusion | 4.102 (8.479)
  IL-6: Day 43: Pre-Infusion: number analyzed (Participants) | 28
  IL-6: Day 43: Pre-Infusion | 1.501 (1.555)
  MCP-1: Day 1: Pre-Infusion | 671.025 (203.263)
  MCP-1: Day 8: 168 hours Post Infusion | 730.466 (284.028)
  MCP-1: Day 43: Pre-Infusion: number analyzed (Participants) | 28
  MCP-1: Day 43: Pre-Infusion | 775.411 (280.839)
  TNF-alpha: Day 1: Pre-Infusion | 3.674 (2.081)
  TNF-alpha: Day 8: 168 hours Post Infusion | 4.475 (4.195)
  TNF-alpha: Day 43: Pre-Infusion: number analyzed (Participants) | 28
  TNF-alpha: Day 43: Pre-Infusion | 3.694 (1.195)
  IL-8: Day 1: Pre-Infusion | 46.254 (43.728)
  IL-8: Day 8: 168 hours Post Infusion | 54.107 (56.734)
  IL-8: Day 43: Pre-Infusion: number analyzed (Participants) | 28
  IL-8: Day 43: Pre-Infusion | 38.674 (30.178)

17. Secondary Outcome: Expansion Cohort: Log Fold Change From Baseline in Cytokine Levels
Description: Cytokine analysis was performed to evaluate levels of Monocyte chemoattractant protein-1 (MCP-1) and various interleukins (including IL-5, IL-6, IL-8), Tumor necrosis factors-alpha (TNF-alpha) and Interferon-gamma (IFN-gamma) in serum samples. Log fold change from baseline (logFC) was defined as logFC (cytokine at time t) = log (cytokine signal at time t) - log (cytokine signal at baseline).
Time Frame: Baseline (Day 1 [Pre-infusion]), Day 8 (168 hour after infusion) and Day 43 (Pre-infusion)
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: log fold change
Arm/Group | Expansion Cohort: Avelumab 10 mg/kg
Number analyzed (Participants) | 40
log fold change
  IFN-gamma: Day 8: 168 hours Post Infusion | 0.697 (1.140)
  IFN-gamma: Day 43: Pre-Infusion: number analyzed (Participants) | 28
  IFN-gamma: Day 43: Pre-Infusion | 0.484 (1.371)
  IL-5: Day 8: 168 hours Post Infusion | 0.080 (1.209)
  IL-5: Day 43: Pre-Infusion: number analyzed (Participants) | 28
  IL-5: Day 43: Pre-Infusion | 0.192 (1.466)
  IL-6: Day 8: 168 hours Post Infusion | 0.476 (2.172)
  IL-6: Day 43: Pre-Infusion: number analyzed (Participants) | 28
  IL-6: Day 43: Pre-Infusion | 0.880 (2.184)
  MCP-1: Day 8: 168 hours Post Infusion | 0.082 (0.353)
  MCP-1: Day 43: Pre-Infusion: number analyzed (Participants) | 28
  MCP-1: Day 43: Pre-Infusion | 0.115 (0.420)
  TNF-alpha: Day 8: 168 hours Post Infusion | 0.209 (0.377)
  TNF-alpha: Day 43: Pre-Infusion: number analyzed (Participants) | 28
  TNF-alpha: Day 43: Pre-Infusion | 0.156 (0.366)
  IL-8: Day 8: 168 hours Post Infusion | 0.199 (0.444)
  IL-8: Day 43: Pre-Infusion: number analyzed (Participants) | 28
  IL-8: Day 43: Pre-Infusion | 0.256 (0.664)

18. Secondary Outcome: Expansion Cohort: Number of Participants With Best Overall Response (BOR) According to Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1
Description: Confirmed BOR was defined as the best response of any of the complete response (CR), partial response (PR), stable disease (SD) and progressive disease (PD) recorded from the date of randomization until disease progression or recurrence (taking the smallest measurement recorded since the start of treatment as reference). CR: Disappearance of all evidence of target and non-target lesions. PR: At least 30% reduction from baseline in the sum of the longest diameter (SLD) of all lesions. SD: Neither sufficient increase to qualify for PD nor sufficient shrinkage to qualify for PR. PD was defined as at least a 20% increase in the SLD, taking as reference the smallest SLD recorded from baseline or the appearance of 1 or more new lesions and unequivocal progression of non-target lesions. Number of participants with best overall response in each category (CR, PR, SD, PD) was reported.
Time Frame: Time from first dose of study treatment up to 1906 days
Population: Safety analysis set included all participants who have received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Expansion Cohort: Avelumab 10 mg/kg
Number analyzed (Participants) | 40
Participants
  Complete response (CR) | 1
  Partial Response (PR) | 3
  Stable disease (SD) | 17
  Progressive disease (PD) | 17
  Non-evaluable (NE) | 2

19. Secondary Outcome: Expansion Cohort: Number of Participants With Immune-related Best Overall Response (irBOR) According to Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1
Description: BOR: best response of any of immune related complete response (irCR), immune related partial response (irPR), immune related stable disease (irSD) and immune related progressive disease (irPD) recorded from the date of randomization until disease progression or recurrence (taking the smallest measurement recorded since the start of treatment as reference). irCR: Complete disappearance of all tumor lesions (both index and non-index lesions with no new measurable/unmeasurable lesions). irPR: At least 30% reduction from baseline in the sum of the longest diameter (SLD) of all lesions). irSD: SLD of target and new measurable lesions neither irCR, irPR, or irPD. irPD: SLD of target and new measurable lesions increases greater than or equal to [>=] 20%, confirmed by a repeat, consecutive observations at least 4 weeks from the date first documented. Number of participants with immune-related best overall response in each category (irCR, irPR, irSD, irPD) was reported.
Time Frame: Time from first dose of study treatment up to 1906 days
Population: Safety analysis set included all participants who have received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Expansion Cohort: Avelumab 10 mg/kg
Number analyzed (Participants) | 40
Participants
  Immune-related Complete response (irCR) | 1
  Immune-related Partial Response (irPR) | 3
  Immune-related Stable disease (irSD) | 21
  Immune-related Progressive disease (irPD) | 9
  Non-evaluable (NE) | 6

20. Secondary Outcome: Expansion Cohort: Progression-Free Survival (PFS) Time According to Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1
Description: PFS was defined as the time from date of randomization until date of the first documentation of progressive disease (PD) or death due to any cause in the absence of documented PD, whichever occurs first. PD was defined as at least a 20 percent (%) increase in the sum of longest diameter (SLD), taking as reference the smallest SLD recorded from baseline or the appearance of 1 or more new lesions and unequivocal progression of non-target lesions. PFS was measured using Kaplan-Meier (KM) estimates.
Time Frame: Time from first dose of study treatment up to 1906 days
Population: Safety analysis set included all participants who have received at least 1 dose of study treatment.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Expansion Cohort: Avelumab 10 mg/kg
Number analyzed (Participants) | 40
weeks | 10.64 [6.00 to 12.00]

21. Secondary Outcome: Expansion Cohort: Immune-related Progression-Free Survival (irPFS) Time According to Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1
Description: irPFS was defined as the time from the first dose of study treatment to the date of first documentation of immune-related progressive disease [irPD] (which was subsequently confirmed) or death due to any cause, whichever occurred first. irPD was defined as the sum of the longest diameters of target and new measurable lesions increases greater than or equal to [>=] 20 percent (%), confirmed by a repeat, consecutive observations at least 4 weeks from the date first documented.
Time Frame: Time from first dose of study treatment up to 1906 days
Population: Safety analysis set included all participants who have received at least 1 dose of study treatment.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Expansion Cohort: Avelumab 10 mg/kg
Number analyzed (Participants) | 40
weeks | 12.00 [10.14 to 12.86]

22. Secondary Outcome: Expansion Cohort: Overall Survival (OS) Time
Description: The OS time was defined as the time from randomization to the date of death. The participants who were still alive at the time of data analysis or who were lost to follow-up OS time was censored at the last recorded date that the participant was known to be alive before the data cutoff date. OS was measured using Kaplan-Meier (KM) estimates.
Time Frame: Time from first dose of study treatment up to 1906 days
Population: Safety analysis set included all participants who have received at least 1 dose of study treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Expansion Cohort: Avelumab 10 mg/kg
Number analyzed (Participants) | 40
months | 8.87 [7.23 to 10.97]

23. Secondary Outcome: Expansion Cohort: Number of Participants With Treatment-Emergent Adverse Events (TEAEs), Serious TEAEs, TEAEs Leading to Death, and TEAEs Leading to Discontinuation
Description: as for outcome 12
Time Frame: Time from first dose of study treatment up to 1906 days
Population: Safety analysis set included all participants who have received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Expansion Cohort: Avelumab 10 mg/kg
Number analyzed (Participants) | 40
Participants
  TEAEs | 40
  Serious TEAEs | 11
  TEAEs Leading to Discontinuation | 7
  TEAEs Leading To Death | 3

24. Secondary Outcome: Expansion Cohort: Number of Participants With Treatment-Emergent Positive Human Anti-Human Antibody (HAHA)
Description: Number of participants with positive HAHA were reported. Participants not having positive HAHA prior to treatment with avelumab and with at least one positive post-baseline result in the HAHA assay were characterized as treatment-emergent. Treatment-emergent participants were further classified as Transient Positive or Persistent positive participants were considered as transient positive if time between first and last positive result was less than 16 weeks apart and a negative result at the most recent visit. Participants were considered as persistent positive if time between first and last positive result >=16 weeks apart or a positive evaluation at the most recent visit.
Time Frame: Day 15 up to Day 1906
Population: Safety analysis set included all participants who have received at least 1 dose of study treatment. Here, "Overall Number of Participants Analyzed" signified participants who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Expansion Cohort: Avelumab 10 mg/kg
Number analyzed (Participants) | 38
Participants
  Transient positive treatment emergent | 2
  Persistent positive treatment emergent | 5

ADVERSE EVENTS:
Time Frame: Dose-escalation Cohort: up to 2205 days and Expansion Cohort: up to 1906 days
Arm/Group | Dose-escalation Cohort: Avelumab 3 mg/kg | Dose-escalation Cohort: Avelumab 10 mg/kg | Dose-escalation Cohort: Avelumab 20 mg/kg | Expansion Cohort: Avelumab 10 mg/kg
All-Cause Mortality (participants affected / at risk) | 4/5 | 3/6 | 4/6 | 36/40
Serious Adverse Events (participants affected / at risk) | 1/5 | 0/6 | 2/6 | 11/40
Other Adverse Events (participants affected / at risk) | 5/5 | 6/6 | 5/6 | 38/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dose-escalation Cohort: Avelumab 3 mg/kg (N=5) | Dose-escalation Cohort: Avelumab 10 mg/kg (N=6) | Dose-escalation Cohort: Avelumab 20 mg/kg (N=6) | Expansion Cohort: Avelumab 10 mg/kg (N=40)
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 1
Biliary tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Disease progression (General disorders) | 1 | 0 | 0 | 2
Multiple organ dysfunction syndrome (General disorders) | 0 | 0 | 0 | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Altered state of consciousness (Nervous system disorders) | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 0
Tonic convulsion (Nervous system disorders) | 0 | 0 | 1 | 0
Platelet count decreased (Investigations) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dose-escalation Cohort: Avelumab 3 mg/kg (N=5) | Dose-escalation Cohort: Avelumab 10 mg/kg (N=6) | Dose-escalation Cohort: Avelumab 20 mg/kg (N=6) | Expansion Cohort: Avelumab 10 mg/kg (N=40)
Vomiting (Gastrointestinal disorders) | 2 | 1 | 2 | 9
Nausea (Gastrointestinal disorders) | 3 | 1 | 0 | 11
Stomatitis (Gastrointestinal disorders) | 1 | 3 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 5
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 3
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 4
Cheilitis (Gastrointestinal disorders) | 0 | 0 | 0 | 3
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Periodontal disease (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 2 | 1 | 7
Non-cardiac chest pain (General disorders) | 1 | 1 | 0 | 0
Fatigue (General disorders) | 0 | 1 | 0 | 5
Influenza like illness (General disorders) | 1 | 0 | 0 | 0
Oedema peripheral (General disorders) | 1 | 0 | 0 | 0
White blood cell count decreased (Investigations) | 1 | 2 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 1 | 0 | 3
Weight decreased (Investigations) | 1 | 1 | 0 | 5
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 1 | 0
Blood creatinine increased (Investigations) | 1 | 0 | 0 | 0
Eosinophil count increased (Investigations) | 0 | 0 | 1 | 0
Neutrophil count decreased (Investigations) | 0 | 1 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 1 | 1 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 1 | 0 | 7
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 5
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 4
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0
Seborrhoea (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Skin atrophy (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 2 | 2 | 5
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 12
Anaemia of malignant disease (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 1 | 1 | 3
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 4
Oral herpes (Infections and infestations) | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 1 | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 3
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 9
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 4
Insomnia (Psychiatric disorders) | 0 | 1 | 1 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Seasonal allergy (Immune system disorders) | 1 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 1 | 1 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 1 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 4
Retinal vein occlusion (Eye disorders) | 0 | 0 | 1 | 0
Visual impairment (Eye disorders) | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 1 | 0 | 0
Hyporthyroidism (Endocrine disorders) | 0 | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 1 | 0
Influenza (Infections and infestations) | 1 | 0 | 0 | 0
Paronychia (Infections and infestations) | 1 | 0 | 0 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Eye discharge (Eye disorders) | 0 | 0 | 1 | 0
Ureterolithiasis (Renal and urinary disorders) | 0 | 1 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 4
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No